CLINICAL TRIAL: NCT01800318
Title: Does Noninvasive Electrical Stimulation of Acupuncture Points (NESAP) Reduce Heelstick Pain in Infants?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 109236
Record Dates: First submitted 2013-02-21; First posted 2013-02-27 (Estimated); Results first posted 2015-12-11 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2017-01

CONDITIONS: Pain
Keywords: NESAP; sucrose; pain; infants
MeSH Terms: conditions — Pain | interventions — Sucrose; Water

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Sham NESAP with 24% oral sucrose (Experimental): 1. Sham NESAP: Four Stim Care electrodes with gel backing will be placed on the infant's lower leg at acupuncture points. However, the Empi Select TENS unit will not be turned on. The TENS unit will be hidden from investigators so that they are blinded to the status of the unit.
  2. Infant will receive 1 ml of 24% oral sucrose solution given along with a pacifier two minutes before the heel stick. Investigators will be blinded to the solution given.
  Interventions: Behavioral: 24% oral Sucrose; Device: Sham NESAP
- NESAP with oral water (Experimental): 1. NESAP: Four Stim Care electrodes with gel backing will be placed on the infant's lower leg at acupuncture points. 10 minutes before the heel stick, the Empi Select TENS unit will be turned on with settings 3.5mA, 10 Hz. The TENS unit will be hidden from investigators so that they are blinded to the status of the unit.
  2. Infant will receive 1 ml of sterile water given via oral syringe along with a pacifier two minutes before the heel stick. Investigators will be blinded to the solution given
  Interventions: Device: NESAP; Behavioral: Oral water
- NESAP with 24% oral sucrose (Experimental): 1. NESAP: Four Stim Care electrodes with gel backing will be placed on the infant's lower leg at acupuncture points. The Empi Select TENS unit will be turned on ten minutes before the heel stick at settings 3.5 mA, 10 Hz. The TENS unit will be hidden from investigators so that they are blinded to the status of the unit.
  2. Infant will receive 1 ml of 24% oral sucrose solution given along with a pacifier two minutes before the heel stick. Investigators will be blinded to the solution given.
  Interventions: Device: NESAP; Behavioral: 24% oral Sucrose
- Sham NESAP with oral water (Placebo Comparator): 1. Sham NESAP: Four Stim Care electrodes with gel backing will be placed on the infant's lower leg at acupuncture points. However, the Empi Select TENS unit will not be turned on. The TENS unit will be hidden from investigators so that they are blinded to the status of the unit.
  2. Infant will receive 1 ml of sterile water given via oral syringe along with a pacifier two minutes before the heel stick. Investigators will be blinded to the solution given.
  Interventions: Device: Sham NESAP; Behavioral: Oral water

INTERVENTIONS:
Device: NESAP — Electrical stimulation will be administered via the Empi Select, a standard TENS unit. To produce analgesia, small electrodes will be placed in treatment groups on the baby's legs at specific acupuncture points: ZuSanLi (ST36), SanYinJiao (SP6), Shen Mai (Bl60), and Shui Quan (KI3)46. StimCare electrodes with a gel base will be applied to the skin ; the skin will not be punctured by these procedures. A low continuous current will be provided with minimal voltage of 3.5 mA. The frequency will be delivered using a stimulation of 10 Hz for 10±1 minutes prior to the heelstick, with continued stimulation during and for 2 minutes after the heel stick. The display will be hidden from view to prevent the rater from being able to observe whether the unit is on.
  Other Names: NESAP using Empi Select TENS unit
  Arms: NESAP with 24% oral sucrose; NESAP with oral water
Behavioral: 24% oral Sucrose — One ml 24% sucrose will be given approximately two minutes before the heel stick. Sucrose will be given via oral syringe along with a pacifier.
  Other Names: Sweet-Ease
  Arms: NESAP with 24% oral sucrose; Sham NESAP with 24% oral sucrose
Device: Sham NESAP — Four electrodes will be placed on the infant's lower leg, but the TENS unit will not be turned on. The TENS unit will be covered and investigators will not know whether the TENS unit is turned on or not (sham NESAP).
  Other Names: Sham NESAP using Empi Select TENS unit
  Arms: Sham NESAP with 24% oral sucrose; Sham NESAP with oral water
Behavioral: Oral water — For infants in the control group, 1 ml of water will be given via oral syringe along with a pacifier 2 minutes before the heel stick. Investigators will be blinded on whether the infants are receiving water or oral sucrose.
  Arms: NESAP with oral water; Sham NESAP with oral water

SUMMARY:
The purpose of the study is to determine whether noninvasive electrical stimulation at acupuncture points (NESAP) and/or 24% sucrose is effective in reducing pain in infants during invasive procedures.

The investigators hypothesize that:

* Gentle noninvasive electrical stimulation at selected acupuncture points and/or oral use of 24% sucrose with pacifier will reduce the newborn infant's responses to heelstick pain, as measured by the Premature Infant Pain Profile (PIPP), heart rate variability, duration of crying, and salivary cortisol levels.
* The effects of combined therapies will be additive.
* The analgesic effects of NESAP and/or sucrose will continue for the duration of the heelstick, reflected by the first two minutes of heelstick and the first two minutes of recovery.

DETAILED DESCRIPTION:
A collaborative prospective, double-blind, randomized trial will be performed at the University of Arkansas for Medical Sciences Hospital (Little Rock, AR), and Lucille Packard Children's Hospital (Palo Alto, CA). After obtaining IRB approval at both sites and parental consent, newborn infants less than 3 days of age who require heelsticks for clinical blood sampling will be randomized in a 2 × 2 factorial trial design to four groups: standard pain management with pacifier and water, Non-invasive Electrical Stimulation of Acupuncture Points (NESAP) with pacifier and water, 24% oral sucrose solution with pacifier, or NESAP plus oral sucrose solution and pacifier prior to their heelstick.

We will study the pain response to the heelstick routinely used to obtain blood for term neonatal infants by enrolling up to 192 infants, 96 from University of Arkansas for Medical Sciences and 96 from Lucille Packard Children's Hospital. This number will allow for screen failures and withdrawals. A minimum of 164 infants collectively from both sites is required to complete the study. Infants will be divided into 4 experimental groups:

1. Group A: Sham (fake electrical stimulation) plus sugar water with pacifier before heelstick.
2. Group B: Electrical stimulation plus water with pacifier before heelstick.
3. Group C: Electrical stimulation plus sugar water with pacifier before heelstick.
4. Group D: Sham (fake electrical stimulation) plus water with pacifier before heelstick.

Electrical stimulation will be applied at appropriate acupuncture points using a very low current for 10 minutes, routine for procedural pain. The response to pain will be assessed using a pain scale, heart rate, heart rate variability and oxygen saturation changes, duration of crying, and changes in salivary cortisol levels.

ELIGIBILITY:
Inclusion Criteria:

* Newborn infants born at 37-42 weeks gestational age
* Less than 3 days of age
* Requiring a heelstick for clinically indicated blood sampling
* Written, informed consent from their parents.

Exclusion Criteria:

* Newborns who have received any analgesic treatment
* Exposed to chronic opiates in utero (excluding opiates given only at the time of delivery) or with a positive drug screen based on review of medical records.
* Current maternal cigarette smoking.
* Infants exposed to birth asphyxia (5-minute Apgar scores of <5 or cord pH <7.0).
* Infants on mechanical ventilation.
* Newborns with suspected or confirmed neuromuscular diseases, congenital anomalies, or sepsis.
* Infants with birth trauma to the lower extremities (bruising or other) or those exposed multiple heelsticks in the previous 24 hours (e.g. requiring frequent glucose or bilirubin measurements).
* Infants born from mothers with drug addiction, diabetes, pre-eclampsia, or systemic inflammatory conditions.
* Abnormal neurological exam
* Congenital heart defects
* Enrollment or participation in other studies
* Dermatologic condition in the area of electrode placement or elsewhere
* Local or systemic infection documented or suspected
* Reasonable known allergy to the gel/adhesive
* Bleeding abnormality
* Connection to other medical equipment or devices that might interfere with the workings or functioning of the transcutaneous electrical nerve stimulation (TENS) unit
* Any condition the investigator determines will put the subject at risk if participating in the study.

Ages: 1 Day to 3 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 162 (Actual)
Dates: Start 2013-03; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard W Hall, M.D., Principal Investigator — University of Arkansas
Locations (2):
- United States (2):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Stanford University, Stanford, California

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of recruitment: 4/10/2013 until 12/31/2014. Types of location: Postpartal/newborn units at University of Arkansas for Medical Sciences and Lucille Packard Childrens Hospital associated with Stanford University.
Pre-assignment Details: All infants enrolled in the study were assigned to groups.
Groups:
- Sham NESAP With 24% Oral Sucrose: 1. Sham NESAP: Four Stim Care electrodes with gel backing will be placed on the infant's lower leg at acupuncture points. However, the Empi Select TENS unit will not be turned on. The TENS unit will be hidden from investigators so that they are blinded to the status of the unit.
  2. Infant will receive 1 ml of 24% oral sucrose solution given along with a pacifier two minutes before the heel stick. Investigators will be blinded to the solution given.
     24% oral Sucrose: One ml 24% sucrose will be given approximately two minutes before the heel stick. Sucrose will be given via oral syringe along with a pacifier.
     Sham NESAP: Four electrodes will be placed on the infant's lower leg, but the TENS unit will not be turned on. The TENS unit will be covered and investigators will not know whether the TENS unit is turned on or not (sham NESAP).
- NESAP With Oral Water: (a) NESAP: Four Stim Care electrodes with gel backing will be placed on the infant's lower leg at acupuncture points. 10 minutes before the heel stick, the Empi Select TENS unit will be turned on. (b) Infant will receive 1 ml of sterile water given via oral syringe along with a pacifier two minutes before the heel stick. Investigators will be blinded to the solution given
  NESAP: Electrical stimulation will be administered via the Empi Select, a standard TENS unit. To produce analgesia, four small electrodes will be placed in treatment groups on the baby's legs at specific acupuncture points. A low continuous current will be provided with minimal voltage of 3.5 mA. The frequency will be delivered using a stimulation of 10 Hz for 10±1 minutes prior to the heelstick, with continued stimulation during and for 2 minutes after the heel stick.
  Oral water:1 ml of water will be given via oral syringe along with a pacifier 2 minutes before the heel stick.
- NESAP With 24% Oral Sucrose: (a) NESAP: Four Stim Care electrodes with gel backing will be placed on the infant's lower leg at acupuncture points. The Empi Select TENS unit will be turned on ten minutes before the heel stick. (b) Infant will receive 1 ml of 24% oral sucrose solution given along with a pacifier two minutes before the heel stick.
  NESAP: Electrical stimulation will be administered via the Empi Select, a standard TENS unit. To produce analgesia, four small electrodes will be placed on the baby's legs at specific acupuncture points. A low continuous current will be provided with minimal voltage of 3.5 mA. The frequency will be delivered using a stimulation of 10 Hz for 10±1 minutes prior to the heelstick, with continued stimulation during and for 2 minutes after the heel stick.
  24% oral Sucrose: One ml 24% sucrose will be given approximately two minutes before the heel stick. Sucrose will be given via oral syringe along with a pacifier.
- Sham NESAP With Oral Water: 1. Sham NESAP: Four Stim Care electrodes with gel backing will be placed on the infant's lower leg at acupuncture points. However, the Empi Select TENS unit will not be turned on. The TENS unit will be hidden from investigators so that they are blinded to the status of the unit.
  2. Infant will receive 1 ml of sterile water given via oral syringe along with a pacifier two minutes before the heel stick. Investigators will be blinded to the solution given.
  Sham NESAP: Four electrodes will be placed on the infant's lower leg, but the TENS unit will not be turned on. The TENS unit will be covered and investigators will not know whether the TENS unit is turned on or not (sham NESAP).
  Oral water: For infants in the control group, 1 ml of water will be given via oral syringe along with a pacifier 2 minutes before the heel stick. Investigators will be blinded on whether the infants are receiving water or oral sucrose.
Period: Overall Study
Arm/Group | Sham NESAP With 24% Oral Sucrose | NESAP With Oral Water | NESAP With 24% Oral Sucrose | Sham NESAP With Oral Water
Started | 39 | 42 | 41 | 40
Completed | 37 | 37 | 40 | 39
Not Completed | 2 | 5 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Newborns randomized to treatment groups during routine newborn screening
Groups:
- NESAP With Oral Water: (a) NESAP: Four Stim Care electrodes with gel backing will be placed on the infant's lower leg at acupuncture points. 10 minutes before the heel stick, the Empi Select TENS unit will be turned on. (b) Infant will receive 1 ml of sterile water given via oral syringe along with a pacifier two minutes before the heel stick.
  NESAP: Electrical stimulation will be administered via the Empi Select, a standard TENS unit. To produce analgesia, four small electrodes will be placed in treatment groups on the baby's legs. at specific acupuncture points. A low continuous current will be provided with minimal voltage of 3.5 mA. The frequency will be delivered using a stimulation of 10 Hz for 10±1 minutes prior to the heelstick, with continued stimulation during and for 2 minutes after the heel stick.
  Oral water: For infants in the control group, 1 ml of water will be given via oral syringe along with a pacifier 2 minutes before the heel stick.
- NESAP With 24% Oral Sucrose: (a) NESAP: Four Stim Care electrodes with gel backing will be placed on the infant's lower leg at acupuncture points. The Empi Select TENS unit will be turned on ten minutes before the heel stick. (b) Infant will receive 1 ml of 24% oral sucrose solution given along with a pacifier two minutes before the heel stick.
  NESAP: Electrical stimulation will be administered via the Empi Select, a standard TENS unit. To produce analgesia, small electrodes will be placed in treatment groups on the baby's legs at four specific acupuncture points. A low continuous current will be provided with minimal voltage of 3.5 mA. The frequency will be delivered using a stimulation of 10 Hz for 10±1 minutes prior to the heelstick, with continued stimulation during and for 2 minutes after the heel stick.
  24% oral Sucrose: One ml 24% sucrose will be given approximately two minutes before the heel stick. Sucrose will be given via oral syringe along with a pacifier.
- Total: Total of all reporting groups
Arm/Group | Sham NESAP With 24% Oral Sucrose | NESAP With Oral Water | NESAP With 24% Oral Sucrose | Sham NESAP With Oral Water | Total
Number analyzed (Participants) | 39 | 42 | 41 | 40 | 162
Age, Continuous [Mean (Standard Deviation); unit: days] | 1 (0.5) | 1 (0.5) | 1 (0.5) | 1 (0.5) | 1 (0.5)
Gender [Count of Participants; unit: Participants]
  Female | 15 | 26 | 16 | 17 | 74
  Male | 24 | 16 | 25 | 23 | 88
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 5 | 7 | 22
  Not Hispanic or Latino | 34 | 37 | 36 | 33 | 140
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 4 | 1 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 12 | 10 | 9 | 19 | 50
  White | 26 | 28 | 29 | 17 | 100
  More than one race | 0 | 0 | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Participants per treatment group [Number; unit: participants] | 39 | 42 | 41 | 40 | 162

OUTCOME MEASURES:

1. Primary Outcome: Changes From Baseline Premature Infant Pain Profile (PIPP) Score to Average PIPP Score During Heel Stick and Squeeze.
Description: The PIPP score includes assessment of contextual, physiological, and behavioral parameters and has been extensively validated for pain assessment in preterm and term infants. PIPP scores were given at baseline before initiation of the TENS unit,and every 30 seconds for the first two minutes of the heel stick and heel squeeze (4 times). The four PIPP scores given during heel stick and squeeze were averaged.
  Behavioral portion of PIPP score: facial expressions are videotaped and analyzed. Physiologic portion of PIPP score: Oxygen saturation levels and heart rates are recorded at baseline and then continuously throughout initiation of the TENS unit and the heel stick procedure. Contextual score - gestational age + sleep/wake state. Subscale scores are added for a total PIPP score. Total or composite PIPP scores are reported.
  Scores on the PIPP for full term infants range from 0-18, with 0 being no pain, 1-6 minimal pain, 7-12 moderate pain, 13-18 severe pain.
Time Frame: Baseline and first two minutes of heel stick an squeeze. PIPP scores are given every 30 seconds for the first two minutes of the heel stick and squeeze and then averaged..
Population: Analysis of PIPP scores assigned during heelstick procedure in newborn infants
Measure: Mean (Standard Deviation); unit: units on a scale (PIPP score)
Arm/Group | Sham NESAP With 24% Oral Sucrose | NESAP With Oral Water | NESAP With 24% Oral Sucrose | Sham NESAP With Oral Water
Number analyzed (Participants) | 37 | 37 | 40 | 39
units on a scale (PIPP score) | 4.0 (1.8) | 5.0 (4.0) | 3.6 (1.2) | 4.9 (4.0)
Statistical Analysis 1: Comparison: Sham NESAP With 24% Oral Sucrose vs NESAP With Oral Water vs NESAP With 24% Oral Sucrose vs Sham NESAP With Oral Water; Test type: Superiority or Other; p = 0.07, ANOVA — RM Anova of effects of treatment groups on PIPP scores:
Statistical Analysis 2: Comparison: Sham NESAP With 24% Oral Sucrose; t test comparing baseline PIPP score with heel stick PIPP scores in group with 24% sucrose and sham NESAP; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; Bonferroni correction
Statistical Analysis 3: Comparison: NESAP With Oral Water; t test comparing baseline PIPP score with heel stick PIPP scores in group with NESAP and oral water; Test type: Superiority or Other; p < 0.01, t-test, 2 sided; Bonferroni correction
Statistical Analysis 4: Comparison: NESAP With 24% Oral Sucrose; t test comparing baseline PIPP score with heel stick PIPP scores in group with 24% sucrose and NESAp combined; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; Bonferroni correction
Statistical Analysis 5: Comparison: Sham NESAP With Oral Water; t test comparing baseline PIPP score with heel stick PIPP scores in standard care group (Sham NESAP with oral water); Test type: Superiority or Other; p < 0.01, t-test, 2 sided; Bonferroni

2. Secondary Outcome: Change in Salivary Cortisol After Heel Stick
Description: Salivary cortisol was obtained prior to initiation of heelstick procedure, and at 5±0.5 minutes after procedure by gentle insertion in the mouth of a soft applicator (Salimetrics Infant Swab). The samples were stored at -20 degrees, and were analyzed at UAMS.
Time Frame: Baseline and 5±0.5 minutes after heel stick
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- NESAP With Oral Water: (a) NESAP: Four Stim Care electrodes with gel backing will be placed on the infant's lower leg at acupuncture points. 10 minutes before the heel stick, the Empi Select TENS unit will be turned on. (b) Infant will receive 1 ml of sterile water given via oral syringe along with a pacifier two minutes before the heel stick.
  NESAP: Electrical stimulation will be administered via the Empi Select, a standard TENS unit. To produce analgesia, small electrodes will be placed in treatment groups on the baby's legs at four specific acupuncture points A low continuous current will be provided with minimal voltage of 3.5 mA. The frequency will be delivered using a stimulation of 10 Hz for 10±1 minutes prior to the heelstick, with continued stimulation during and for 2 minutes after the heel stick.
  Oral water: For infants in the control group, 1 ml of water will be given via oral syringe along with a pacifier 2 minutes before the heel stick.
- NESAP With 24% Oral Sucrose: (a) NESAP: Four Stim Care electrodes with gel backing will be placed on the infant's lower leg at acupuncture points. The Empi Select TENS unit will be turned on ten minutes before the heel stick. (b) Infant will receive 1 ml of 24% oral sucrose solution given along with a pacifier two minutes before the heel stick. NESAP: Electrical stimulation will be administered via the Empi Select, a standard TENS unit. To produce analgesia, small electrodes will be placed in treatment groups on the baby's legs at four specific acupuncture points A low continuous current will be provided with minimal voltage of 3.5 mA. The frequency will be delivered using a stimulation of 10 Hz for 10±1 minutes prior to the heelstick, with continued stimulation during and for 2 minutes after the heel stick.
  24% oral Sucrose: One ml 24% sucrose will be given approximately two minutes before the heel stick. Sucrose will be given via oral syringe along with a pacifier.
Arm/Group | Sham NESAP With 24% Oral Sucrose | NESAP With Oral Water | NESAP With 24% Oral Sucrose | Sham NESAP With Oral Water
Number analyzed (Participants) | 21 | 18 | 20 | 16
ng/ml | 36.6 (28.9) | 41.7 (26) | 58.5 (22) | 56.3 (35.7)
Statistical Analysis 1: Comparison: Sham NESAP With 24% Oral Sucrose vs NESAP With Oral Water vs NESAP With 24% Oral Sucrose vs Sham NESAP With Oral Water; Test type: Superiority or Other; p = 0.9, ANOVA

3. Secondary Outcome: Change in Heart Rate Variability During Heel Stick
Description: Changes in Heart Rate Variability (HRV) were evaluated using the DL 900 monitor with 3-channel output with 5 leads. Premature infant leads from Braemar, Incorporated, were used with the DL 900 monitor. Leads were applied to the infant's chest before initiation of the TENS unit and the heel stick. The DL300 Holter Monitor will started recording HRV within 10 minutes of TENS unit initiation and the heel stick procedure and continued recording during the procedure and for 2 minutes afterwards.
Time Frame: Baseline, 20 minutes +/- 5 minutes
Population: Newborn infants
Measure: Mean (Standard Deviation); unit: LF/HF ratio
Arm/Group | Sham NESAP With 24% Oral Sucrose | NESAP With Oral Water | NESAP With 24% Oral Sucrose | Sham NESAP With Oral Water
Number analyzed (Participants) | 37 | 38 | 40 | 39
LF/HF ratio | 1.4 (1.2) | 1.5 (2) | 1.3 (1.2) | 1.3 (1.4)
Statistical Analysis 1: Comparison: Sham NESAP With 24% Oral Sucrose vs NESAP With Oral Water vs NESAP With 24% Oral Sucrose vs Sham NESAP With Oral Water; Test type: Superiority or Other; p = 0.9, ANOVA

4. Secondary Outcome: Duration of Crying After TENS Unit Was Initiated But Before Heel Stick.
Description: (a) Any crying after initiation of TENS unit was noted. If the PIPP scores increased by 4 points from baseline, the TENS unit would have been turned off and the infant withdrawn from the study (safety outcome).
Time Frame: 10 minutes
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- NESAP With Oral Water: (a) NESAP: Four Stim Care electrodes with gel backing will be placed on the infant's lower leg at acupuncture points. 10 minutes before the heel stick, the Empi Select TENS unit will be turned on. .(b) Infant will receive 1 ml of sterile water given via oral syringe along with a pacifier two minutes before the heel stick. .
  NESAP: Electrical stimulation will be administered via the Empi Select, a standard TENS unit. To produce analgesia, small electrodes will be placed in treatment groups on the baby's legs at four specific acupuncture points. A low continuous current will be provided with minimal voltage of 3.5 mA. The frequency will be delivered using a stimulation of 10 Hz for 10±1 minutes prior to the heelstick, with continued stimulation during and for 2 minutes after the heel stick.
  Oral water: For infants in the control group, 1 ml of water will be given via oral syringe along with a pacifier 2 minutes before the heel stick.
- NESAP With 24% Oral Sucrose: (a) NESAP: Four Stim Care electrodes with gel backing will be placed on the infant's lower leg at acupuncture points. The Empi Select TENS unit will be turned on ten minutes before the heel stick. (b) Infant will receive 1 ml of 24% oral sucrose solution given along with a pacifier two minutes before the heel stick.
  NESAP: Electrical stimulation will be administered via the Empi Select, a standard TENS unit. To produce analgesia, small electrodes will be placed in treatment groups on the baby's legs at four specific acupuncture points A low continuous current will be provided with minimal voltage of 3.5 mA. The frequency will be delivered using a stimulation of 10 Hz for 10±1 minutes prior to the heelstick, with continued stimulation during and for 2 minutes after the heel stick.
  24% oral Sucrose: One ml 24% sucrose will be given approximately two minutes before the heel stick. .
Arm/Group | Sham NESAP With 24% Oral Sucrose | NESAP With Oral Water | NESAP With 24% Oral Sucrose | Sham NESAP With Oral Water
Number analyzed (Participants) | 37 | 37 | 40 | 39
seconds | 0 (0) | 0 (0) | 0 (0) | 0 (0)

5. Secondary Outcome: Duration of Crying During Heel Stick
Description: Any crying during the heel stick procedure was timed in seconds.
Time Frame: 5 minutes +/- 2 minutes
Population: Newborn infants during heel stick procedure, crying timed in seconds
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Sham NESAP With 24% Oral Sucrose | NESAP With Oral Water | NESAP With 24% Oral Sucrose | Sham NESAP With Oral Water
Number analyzed (Participants) | 37 | 37 | 40 | 39
seconds | 0.43 (1.7) | 32 (59.8) | 7.28 (26.9) | 23.7 (57.8)
Statistical Analysis 1: Comparison: Sham NESAP With 24% Oral Sucrose vs NESAP With Oral Water vs NESAP With 24% Oral Sucrose vs Sham NESAP With Oral Water; Test type: Superiority or Other; p = 0.008, ANOVA; F4.048

ADVERSE EVENTS:
Time Frame: 1 year, 8 months
Description: No adverse events. Infants were monitored continuously throughout data collection period using heart monitor, oxygen saturation monitor, facial videotaping, neonatologist present at all times, pediatric physical therapist and nurse practitioner present at all times.
Arm/Group | Sham NESAP With 24% Oral Sucrose | NESAP With Oral Water | NESAP With 24% Oral Sucrose | Sham NESAP With Oral Water
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/37 | 0/40 | 0/39
Other Adverse Events (participants affected / at risk) | 0/37 | 0/37 | 0/40 | 0/39

LIMITATIONS AND CAVEATS:
We had difficulty collecting adequate saliva for salivary cortisol analysis. Many infants had insufficient saliva to run a reliable analysis, and numbers of infants with adequate saliva samples both before and after the heel stick were limited.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes